CLINICAL TRIAL: NCT02562768
Title: Multiple-Ascending Dose, Safety, Tolerability, and Pharmacokinetic Study of LY3154207 in Healthy Subjects and Subjects With Parkinson's Disease
Brief Title: A Study of LY3154207 in Healthy Participants and Participants With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15512; I7S-EW-HBEC (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — LY3154207

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY3154207 (Experimental): LY3154207 administered orally once daily in multiple-ascending dose cohorts for 14 days.
  Interventions: Drug: LY3154207
- Placebo (Placebo Comparator): Placebo matching LY3154207 administered once daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3154207 — Administered orally
  Arms: LY3154207
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
This two-part study will evaluate how safe LY3154207 is and the effects it has on the body.

Part A will include healthy participants. Each participant will receive daily doses of LY3154207 or placebo for 14 days. Part A will last approximately 4 weeks including a 17 day stay in the clinical research unit (CRU) and follow-up.

Part B is contingent on the results of Part A. Part B will include participants with Parkinson's disease. Each participant will receive daily doses of LY3154207 or placebo for 14 days. Part B will last approximately 4 weeks including a 17 day stay in the CRU and follow-up.

Both Part A and Part B will require screening within 30 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Overtly healthy males or females, as determined by medical history and physical examination
* Female participants not of child-bearing potential

Part B:

* Have a clinical diagnosis of idiopathic Parkinson's disease for at least 1 year and on stable medication for at least 4 weeks

Part A and B

* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent
* Have a body mass index (BMI) of 18.0 to 29.9 kilograms per square meter (kg/m²)

Exclusion Criteria:

* Have participated, in the last 30 days, in a clinical trial involving an investigational product
* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs; or constituting a risk when taking the study medication; or interfering with the interpretation of study data

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through study completion (Day 15) in each part.

SECONDARY OUTCOMES:
Plasma (blood) Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY3154207 | At multiple time points from baseline through day 15 in each part
Plasma (blood) Pharmacokinetics: Maximum Concentration (Cmax) of LY3154207 | At multiple time points from baseline through day 15 in each part
Plasma (blood) Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY3154207 after a High-Calorie Meal | Baseline through 24 hours after administration of study drug on Day 10 in Part A.
Plasma (blood) Pharmacokinetics: Maximum Concentration (Cmax) of LY3154207 after a High-Calorie Meal | Baseline through 24 hours after administration of study drug on Day 10 in Part A.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Parexel International LLC, Glendale, California
  - Compass Research, Orlanda, Florida
  - Compass Research, The Villages, Florida

REFERENCES:
- [Derived] Wilbraham D, Biglan KM, Svensson KA, Tsai M, Pugh M, Ardayfio P, Kielbasa W. Safety, Tolerability, and Pharmacokinetics of Mevidalen (LY3154207), a Centrally Acting Dopamine D1 Receptor-Positive Allosteric Modulator, in Patients With Parkinson Disease. Clin Pharmacol Drug Dev. 2022 Mar;11(3):324-332. doi: 10.1002/cpdd.1039. Epub 2021 Oct 19. PMID 34664427
- [Derived] Wilbraham D, Biglan KM, Svensson KA, Tsai M, Kielbasa W. Safety, Tolerability, and Pharmacokinetics of Mevidalen (LY3154207), a Centrally Acting Dopamine D1 Receptor-Positive Allosteric Modulator (D1PAM), in Healthy Subjects. Clin Pharmacol Drug Dev. 2021 Apr;10(4):393-403. doi: 10.1002/cpdd.874. Epub 2020 Oct 7. PMID 33029934
- See also: Click here for more information about this study: A Study of LY3154207 in Participants With Parkinson's Disease (Part B) — http://www.lillytrialguide.com/en-US/studies/parkinson's-disease/HBEC#?postal=